CLINICAL TRIAL: NCT04316884
Title: Uppsala Intensive Care Study of Mechanisms for Organ Dysfunction in Covid-19
Brief Title: Mechanisms for Organ Dysfunction in Covid-19
Acronym: UMODCOVID19
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Robert Frithiof, Associate Professor, Uppsala University
Other Study IDs: EPN 2017/043 Covid19
Record Dates: First submitted 2020-03-13; First posted 2020-03-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: COVID-19; Organ Dysfunction Syndrome Sepsis; Organ Dysfunction Syndrome, Multiple; Septic Shock; Acute Kidney Injury; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Toxemia; Multiple Organ Failure; Shock, Septic; Acute Kidney Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine and Sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19: Patients with suspected or verified COVID-19 admitted to intensive care at Uppsala University Hospital

SUMMARY:
The study aims to investigate organ dysfunction and biomarkers in patients with suspected or verified COVID-19 during intensive care at Uppsala University Hospital.

DETAILED DESCRIPTION:
Consenting patients with suspected or verified SARS-COV-2 infection, COVID-19, will undergo daily blood, urine and sputum sampling during their stay in intensive care. Data on organ dysfunction will be collected through the electronic patient journal and electronic patient data management system. The collected samples will be analysed for a panel of potential biomarkers that will be correlated to organ dysfunction and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to intensive care
* suspected or verified COVID-19

Exclusion Criteria:

* Pregnancy or breastfeeding
* Under-age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients requiring intensive care with suspected or verified COVID19
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | During Intensive Care, an estimated average of 10 days.
  KDIGO AKI score

SECONDARY OUTCOMES:
ARDS | During intensive care, an estimated average of 10 days.
  Acute Respiratory Distress Syndrome yes/no
30 day mortality | 30 days
  Death within 30 days of ICU admission
1 year mortality | 1 year
  Death within 1 year of ICU admission
Chronic Kidney Disease | 60 days and 1 year after ICU admission
  Development of Chronic Kidney Disease
SOFA-score | During Intensive Care, an estimated average of 10 days.
  Sequential Organ Failure Score as a continuous variable
Thromboembolic events | During intensive care
  Occurence of thrombosis and/or embolous
ICUAW | During intensive care or after intensive care
  Intensive care acquired weakness

CONTACTS AND LOCATIONS:
Overall Officials: Robert Frithiof, MD. PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be made available upon reasonable request.

REFERENCES:
- [Result] Hultstrom M, von Seth M, Frithiof R. Hyperreninemia and low total body water may contribute to acute kidney injury in COVID-19 patients in intensive care. J Hypertens. 2020 Aug;38(8):1613-1614. doi: 10.1097/HJH.0000000000002531. No abstract available. PMID 32472780
- [Result] Hultstrom M, Persson B, Eriksson O, Lipcsey M, Frithiof R, Nilsson B. Blood type A associates with critical COVID-19 and death in a Swedish cohort. Crit Care. 2020 Aug 12;24(1):496. doi: 10.1186/s13054-020-03223-8. No abstract available. PMID 32787887
- [Result] Eriksson O, Hultstrom M, Persson B, Lipcsey M, Ekdahl KN, Nilsson B, Frithiof R. Mannose-Binding Lectin is Associated with Thrombosis and Coagulopathy in Critically Ill COVID-19 Patients. Thromb Haemost. 2020 Dec;120(12):1720-1724. doi: 10.1055/s-0040-1715835. Epub 2020 Sep 1. PMID 32871607
- [Result] Stattin K, Lipcsey M, Andersson H, Ponten E, Bulow Anderberg S, Gradin A, Larsson A, Lubenow N, von Seth M, Rubertsson S, Hultstrom M, Frithiof R. Inadequate prophylactic effect of low-molecular weight heparin in critically ill COVID-19 patients. J Crit Care. 2020 Dec;60:249-252. doi: 10.1016/j.jcrc.2020.08.026. Epub 2020 Sep 3. PMID 32920503
- [Result] Frithiof R, Bergqvist A, Jarhult JD, Lipcsey M, Hultstrom M. Presence of SARS-CoV-2 in urine is rare and not associated with acute kidney injury in critically ill COVID-19 patients. Crit Care. 2020 Sep 29;24(1):587. doi: 10.1186/s13054-020-03302-w. No abstract available. PMID 32993742
- [Result] Asif S, Frithiof R, Lipcsey M, Kristensen B, Alving K, Hultstrom M. Weak anti-SARS-CoV-2 antibody response is associated with mortality in a Swedish cohort of COVID-19 patients in critical care. Crit Care. 2020 Nov 6;24(1):639. doi: 10.1186/s13054-020-03362-y. No abstract available. PMID 33158455
- [Result] Luther T, Bulow-Anderberg S, Larsson A, Rubertsson S, Lipcsey M, Frithiof R, Hultstrom M. COVID-19 patients in intensive care develop predominantly oliguric acute kidney injury. Acta Anaesthesiol Scand. 2021 Mar;65(3):364-372. doi: 10.1111/aas.13746. Epub 2020 Nov 28. PMID 33190222
- [Result] Bulow Anderberg S, Luther T, Berglund M, Larsson R, Rubertsson S, Lipcsey M, Larsson A, Frithiof R, Hultstrom M. Increased levels of plasma cytokines and correlations to organ failure and 30-day mortality in critically ill Covid-19 patients. Cytokine. 2021 Feb;138:155389. doi: 10.1016/j.cyto.2020.155389. Epub 2020 Dec 14. PMID 33348065
- [Result] Zhou S, Butler-Laporte G, Nakanishi T, Morrison DR, Afilalo J, Afilalo M, Laurent L, Pietzner M, Kerrison N, Zhao K, Brunet-Ratnasingham E, Henry D, Kimchi N, Afrasiabi Z, Rezk N, Bouab M, Petitjean L, Guzman C, Xue X, Tselios C, Vulesevic B, Adeleye O, Abdullah T, Almamlouk N, Chen Y, Chasse M, Durand M, Paterson C, Normark J, Frithiof R, Lipcsey M, Hultstrom M, Greenwood CMT, Zeberg H, Langenberg C, Thysell E, Pollak M, Mooser V, Forgetta V, Kaufmann DE, Richards JB. A Neanderthal OAS1 isoform protects individuals of European ancestry against COVID-19 susceptibility and severity. Nat Med. 2021 Apr;27(4):659-667. doi: 10.1038/s41591-021-01281-1. Epub 2021 Feb 25. PMID 33633408
- [Result] Lipcsey M, Persson B, Eriksson O, Blom AM, Fromell K, Hultstrom M, Huber-Lang M, Ekdahl KN, Frithiof R, Nilsson B. The Outcome of Critically Ill COVID-19 Patients Is Linked to Thromboinflammation Dominated by the Kallikrein/Kinin System. Front Immunol. 2021 Feb 22;12:627579. doi: 10.3389/fimmu.2021.627579. eCollection 2021. PMID 33692801
- [Result] Jarhult JD, Hultstrom M, Bergqvist A, Frithiof R, Lipcsey M. The impact of viremia on organ failure, biomarkers and mortality in a Swedish cohort of critically ill COVID-19 patients. Sci Rep. 2021 Mar 30;11(1):7163. doi: 10.1038/s41598-021-86500-y. PMID 33785784
- [Result] Frithiof R, Rostami E, Kumlien E, Virhammar J, Fallmar D, Hultstrom M, Lipcsey M, Ashton N, Blennow K, Zetterberg H, Punga AR. Critical illness polyneuropathy, myopathy and neuronal biomarkers in COVID-19 patients: A prospective study. Clin Neurophysiol. 2021 Jul;132(7):1733-1740. doi: 10.1016/j.clinph.2021.03.016. Epub 2021 Apr 1. PMID 33875374
- [Result] Galien S, Hultstrom M, Lipcsey M, Stattin K, Frithiof R, Rosen J; Uppsala Intensive Care COVID-19 Research Group. Point of care ultrasound screening for deep vein thrombosis in critically ill COVID-19 patients, an observational study. Thromb J. 2021 Jun 2;19(1):38. doi: 10.1186/s12959-021-00272-z. PMID 34078399
- [Result] Gradin A, Andersson H, Luther T, Anderberg SB, Rubertsson S, Lipcsey M, Aberg M, Larsson A, Frithiof R, Hultstrom M. Urinary cytokines correlate with acute kidney injury in critically ill COVID-19 patients. Cytokine. 2021 Oct;146:155589. doi: 10.1016/j.cyto.2021.155589. Epub 2021 May 24. PMID 34161857
- [Result] Huckriede J, Anderberg SB, Morales A, de Vries F, Hultstrom M, Bergqvist A, Ortiz-Perez JT, Sels JW, Wichapong K, Lipcsey M, van de Poll M, Larsson A, Luther T, Reutelingsperger C, de Frutos PG, Frithiof R, Nicolaes GAF. Evolution of NETosis markers and DAMPs have prognostic value in critically ill COVID-19 patients. Sci Rep. 2021 Aug 3;11(1):15701. doi: 10.1038/s41598-021-95209-x. PMID 34344929
- [Result] Pellegrini M, Larina A, Mourtos E, Frithiof R, Lipcsey M, Hultstrom M, Segelsjo M, Hansen T, Perchiazzi G. A quantitative analysis of extension and distribution of lung injury in COVID-19: a prospective study based on chest computed tomography. Crit Care. 2021 Aug 4;25(1):276. doi: 10.1186/s13054-021-03685-4. PMID 34348797
- [Result] Karawajczyk M, Douhan Hakansson L, Lipcsey M, Hultstrom M, Pauksens K, Frithiof R, Larsson A. High expression of neutrophil and monocyte CD64 with simultaneous lack of upregulation of adhesion receptors CD11b, CD162, CD15, CD65 on neutrophils in severe COVID-19. Ther Adv Infect Dis. 2021 Jul 31;8:20499361211034065. doi: 10.1177/20499361211034065. eCollection 2021 Jan-Dec. PMID 34377464
- [Result] Huckriede J, de Vries F, Hultstrom M, Wichapong K, Reutelingsperger C, Lipcsey M, Garcia de Frutos P, Frithiof R, Nicolaes GAF. Histone H3 Cleavage in Severe COVID-19 ICU Patients. Front Cell Infect Microbiol. 2021 Sep 10;11:694186. doi: 10.3389/fcimb.2021.694186. eCollection 2021. PMID 34568088
- [Result] Bulow Anderberg S, Lipcsey M, Hultstrom M, Eriksson AK, Venge P, Frithiof R, On Behalf Of The Uppsala Intensive Care Covid-Research Group. Systemic Human Neutrophil Lipocalin Associates with Severe Acute Kidney Injury in SARS-CoV-2 Pneumonia. J Clin Med. 2021 Sep 14;10(18):4144. doi: 10.3390/jcm10184144. PMID 34575252
- [Result] Sancho Ferrando E, Hanslin K, Hultstrom M, Larsson A, Frithiof R, Lipcsey M; Uppsala Intensive Care COVID-19 Research Group. Soluble TNF receptors predict acute kidney injury and mortality in critically ill COVID-19 patients: A prospective observational study. Cytokine. 2022 Jan;149:155727. doi: 10.1016/j.cyto.2021.155727. Epub 2021 Oct 5. PMID 34628127
- [Result] Nakanishi T, Pigazzini S, Degenhardt F, Cordioli M, Butler-Laporte G, Maya-Miles D, Bujanda L, Bouysran Y, Niemi ME, Palom A, Ellinghaus D, Khan A, Martinez-Bueno M, Rolker S, Amitrano S, Roade Tato L, Fava F; FinnGen; COVID-19 Host Genetics Initiative (HGI); Spinner CD, Prati D, Bernardo D, Garcia F, Darcis G, Fernandez-Cadenas I, Holter JC, Banales JM, Frithiof R, Kiryluk K, Duga S, Asselta R, Pereira AC, Romero-Gomez M, Nafria-Jimenez B, Hov JR, Migeotte I, Renieri A, Planas AM, Ludwig KU, Buti M, Rahmouni S, Alarcon-Riquelme ME, Schulte EC, Franke A, Karlsen TH, Valenti L, Zeberg H, Richards JB, Ganna A. Age-dependent impact of the major common genetic risk factor for COVID-19 on severity and mortality. J Clin Invest. 2021 Dec 1;131(23):e152386. doi: 10.1172/JCI152386. PMID 34597274
- [Result] COVID-19 Host Genetics Initiative. Mapping the human genetic architecture of COVID-19. Nature. 2021 Dec;600(7889):472-477. doi: 10.1038/s41586-021-03767-x. Epub 2021 Jul 8. PMID 34237774
- [Derived] Bjarnadottir KJ, Perchiazzi G, Sidenbladh CL, Larina A, Wallin E, Larsson IM, Franzen S, Larsson AO, Sousa MLA, Segelsjo M, Hansen T, Frithiof R, Hultstrom M, Lipcsey M, Pellegrini M. Body mass index is associated with pulmonary gas and blood distribution mismatch in COVID-19 acute respiratory failure. A physiological study. Front Physiol. 2024 Jul 10;15:1399407. doi: 10.3389/fphys.2024.1399407. eCollection 2024. PMID 39050483
- [Derived] Halvorsen P, Hultstrom M, Hastbacka J, Larsson IM, Eklund R, Arnberg FK, Hokkanen L, Frithiof R, Wallin E, Orwelius L, Lipcsey M. Health-related quality of life after surviving intensive care for COVID-19: a prospective multicenter cohort study. Sci Rep. 2023 Oct 21;13(1):18035. doi: 10.1038/s41598-023-45346-2. PMID 37865685
- [Derived] Bark L, Larsson IM, Wallin E, Simren J, Zetterberg H, Lipcsey M, Frithiof R, Rostami E, Hultstrom M. Central nervous system biomarkers GFAp and NfL associate with post-acute cognitive impairment and fatigue following critical COVID-19. Sci Rep. 2023 Aug 12;13(1):13144. doi: 10.1038/s41598-023-39698-y. PMID 37573366
- [Derived] Perchiazzi G, Larina A, Hansen T, Frithiof R, Hultstrom M, Lipcsey M, Pellegrini M. Chest dual-energy CT to assess the effects of steroids on lung function in severe COVID-19 patients. Crit Care. 2022 Oct 25;26(1):328. doi: 10.1186/s13054-022-04200-z. PMID 36284360
- [Derived] Hultstrom M, Lipcsey M, Morrison DR, Nakanishi T, Butler-Laporte G, Chen Y, Yoshiji S, Forgetta V, Farjoun Y, Wallin E, Larsson IM, Larsson A, Marton A, Titze JM, Nihlen S, Richards JB, Frithiof R. Dehydration is associated with production of organic osmolytes and predicts physical long-term symptoms after COVID-19: a multicenter cohort study. Crit Care. 2022 Oct 21;26(1):322. doi: 10.1186/s13054-022-04203-w. PMID 36271419